CLINICAL TRIAL: NCT02749448
Title: The Effect of Autologous Adipose Mesenchymal Stem Cells in Treatment of Airway Injury in Patients Exposed to Sulfur Mustard
Brief Title: Mesenchymal Stem Cells Therapy for Treatment of Airway Remodeling in Mustard Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Mostafa Ghanei (Other)
Responsible Party: Sponsor-Investigator, Dr. Mostafa Ghanei, pulmonologist doctor, Baqiyatallah Medical Sciences University
Organization: Baqiyatallah Medical Sciences University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCT2015110524890N1
Record Dates: First submitted 2016-04-09; First posted 2016-04-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mesenchymal stem cell (Other): There are complex sets of non-hematopoietic cells in bone marrow called mesenchymal progenitor cells (MPCs). MSCs are well-known as multipotent cells that have the ability to self-renew and differentiate into a great variety of cells. MSCs can be isolated from bone marrow, umbilical cord, peripheral blood and adipose tissue, and cultured in specific media. MSC colony formation, which is known as marrow-like stromal cells and MPCs, is similar to fibroblast colony forming unit (CFU-F) in in vitro condition. According to the International Society for Cellular Therapy (ISCT), MSCs can be easily detected or identified from other cells using flow cytometric analysis to detect specific surface markers
  Interventions: Other: mesenchymal stem cell

INTERVENTIONS:
Other: mesenchymal stem cell — There are complex sets of non-hematopoietic cells in bone marrow called mesenchymal progenitor cells (MPCs). MSCs are well-known as multipotent cells that have the ability to self-renew and differentiate into a great variety of cells. MSCs can be isolated from bone marrow, umbilical cord, peripheral blood and adipose tissue, and cultured in specific media. MSC colony formation, which is known as marrow-like stromal cells and MPCs, is similar to fibroblast colony forming unit (CFU-F) in in vitro condition. According to the International Society for Cellular Therapy (ISCT), MSCs can be easily detected or identified from other cells using flow cytometric analysis to detect specific surface markers

SUMMARY:
Background: Sulfur mustard (SM) is a potent alkylating agent that targets several organs, especially lung tissue. SM exposure leads to serious changes in morphological structure of airway system, which is associated with chronic obstructive pulmonary deficiency following exposure to SM. With extensive progress and achievements in tissue repair through stem cells therapy, consideration of lung tissue has been increased due to the high prevalence of pulmonary problems. Several factors such as selection of cell types, required conditions for growth and proliferation of stem cells, and the process of entering into the body to repair damaged lung tissue are considered as the most important problems in this issue. Accumulating studies, both in animals and human with mesenchymal stem cells (MSC) support the hypothesis of therapeutic effects of these cells in various disorders. In this study investigators aimed to evaluate safety and potential efficacy of systemic MSC administration for treatment of chronic lung injuries in SM-exposed patients.

Methods: Patients will receive 100 million MSC cells every two months for three injections within 6 months. After each injection, parameters including safety, pulmonary function testing (PFT), quality-of-life indicators, 6 minute walk test (6MWT), and expression of inflammation and oxidative stress genes will be evaluated.

DETAILED DESCRIPTION:
Patients selection:

In this clinical trial, investigators considered therapeutic effect of MSCs in SM-exposed male patients.Patients, had a documented encounter with SM during the Iran-Iraq war. The patients signed informed consent before study. They were selected according to the following criteria: (a) the severity of lung injury was ranged from moderate 50< forced expiratory volume in 1 second (FEV1) <65 to severe 40<FEV1<50; (b) absence of contraindications spirometry (hemoptysis, cerebral arterial aneurysm or aortic, pulmonary embolism, uncontrolled blood pressure, recent pneumothorax, no doubt surgery/thoracic recent, recent stroke); and (c) no coagulation. The exclusion criteria for the selection process were as follow: (a) participate in another study at the same time; (b) smoking habitat; (c) the existence of pneumonia during the study; (d) the incidence of transfusion reaction; (e) underlying other diseases (cardiovascular disease, hypertension, diabetes).

Isolation and culture of adipose derived stem cells:

200mL of abdominal adipose tissue was obtained under local anesthesia by liposuction aspirates protocol. The lipoaspirate was washed with PBS to remove tissue debris. 100mL PBS containing 0.1% w/v collagenase A type I was added to isolated tissue and then incubated at 37ºC for 60 minutes. Collagenase activity was neutralized using MEM medium along with 10% fetal bovine serum. Cell pellets were resuspended in culture medium after centrifugation at 2000rpm for 10 min, and then transferred to culture flasks for 72 h at 37ºC in 5% CO2 condition. The culture medium in the flasks was changed every 3 days, and cells were passaged for two times.

Flow cytometry analysis:

To analyze the cell surface antigen expression, 5×105 fresh cells from third passage were harvested by trypsin-EDTA. Cells were centrifuged at 100 g for 1 min, resuspended in stain buffer (PBS, 2% FBS) and then incubated on ice for 10 minutes. Trypsin was neutralized by centrifuge and isolated cells were washed twice with PBS and finally resuspended in stain buffer. Cells were incubated in dark environment for 30 minutes. After incubation, the cells were labeled with anti-human monoclonal antibodies (MAbs) conjugated to fluorochromes. These antibodies were as follow: anti-CD90-fluorescein isothiocyanate (FITC), CD73-phycoerythrin (PE), CD11b-FITC, CD34-FITC, CD44-FITC, CD45-PE, CD105-PE. The frequencies of all immunolabeled cells were analyzed by FACS Canto II flow cytometer, in which approximately 500,000 events were assessed and data were analyzed using FlowJo software (version 10.0).

Karyotype analysis for abnormalities detection:

Standard Giemsa staining procedure was performed and chromosome preparations were obtained from 80% confluent cells. To stop microtubule formation, the cells were treated with Colcemid solution. The mitotic arrested cells were then harvested using trypsin-EDTA. The cells were extracted and then immersed in 75 mmol/l KCl for 30 minute at laboratory temperature. Finally, they obtained by a centrifugation. The supernatant was replaced with fixative solution and the suspension was spread over slides for microscopic examination and imaging. At least, 15 metaphase spreads were analyzed. The karyotypes were considered with light microscope using a cytovision software.

Freezing and Storage of Adipose-derived Stem Cells:

ADMSCs were harvested at 90% confluence before injection for freezing. To collect cells, culture medium was removed and replaced with sterile PBS and after three minutes it was replaced with trypsin-EDTA solution and then incubated at 37°C for 5 minutes. Complete medium (MEM with 10% FBS) was added to inactivate the trypsin, and centrifuged at 1500 rpm for 5 minutes. Cell pellet was resuspended in cryopreservation medium (80% FBS, 10% dimethylsulfoxide and 10% MEM medium) with a final concentration of 5 million cells per milliliter and aliquoted into cryovials. The vials stored at -80 °C overnight and then transferred into a liquid nitrogen container for long-term storage.

MSCs injection and Study plan:

Patients received 100×106 cells every 20 day for four injections within 2 months and screened for 7 times. MSCs were injected intravenously along with 300 ml normal saline to the patient at a maximum rate of 2×106 cells/min. Each infusion took approximately 30 minute to be completed. After each injection, patient stayed at hospital for at least 6h as recovery time. Efficacy of MSCs treatment in these patients were evaluated using the following parameters: pulmonary functions test (PFTs) [forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC), FEV1/FVC], total lung capacity by body plethysmography, single-breath carbon monoxide diffusing capacity (CO diffusion) , exercise performance [6-minute walk test (6MWT)], Borg scale dyspnea assessment (BSDA), COPD Assessment Test (CAT), St. George's Respiratory Questionnaire (SRGQ) and comprehensive safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients who had a documentary exposure to mustard gas in the Iran-Iraq war
* their disease severity were as following based on spirometric: moderate 50<forced expiratory volume at one second (FEV1)<65 or severe 40<FEV1<50
* absence of contraindications spirometry (recent myocardial ischemia (MI)
* hemoptysis
* cerebral arterial aneurysm or aortic
* pulmonary embolism,
* uncontrolled blood pressure
* recent pneumothorax
* no doubt surgery/recent thoracic
* recent eye surgery, recent stroke
* non-availability in another research study at a same time
* no coagulation disorders

Exclusion Criteria:

* smoking
* the incidence of pneumonia during the study
* the incidence of transfusion reaction
* other medical condition (cardiovascular disease, hypertension, diabetes)
* visiting less than 2 times

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
pulmonary function testing (PFT) | one year
  Pulmonary Function Testing (PFT) is a complete evaluation of the respiratory system including patient history, physical examinations, chest x-ray examinations, arterial blood gas analysis, and tests of pulmonary function. The primary purpose of pulmonary function testing is to identify the severity of pulmonary impairment.

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | one year
  The SGRQ is designed to measure health impairment in patients with asthma and COPD. It is also valid for use in bronchiectasis and has been used successfully in SM patients
6 minute walk test (6MWT) | one year
  The original purpose of the six minute walk was to test exercise tolerance in chronic respiratory disease and heart failure.

IPD SHARING:
Plan to Share IPD: No
there is no individual participant data

REFERENCES:
- [Derived] Marzouni ET, Dorcheh SP, Nejad-Moghaddam A, Ghanei M, Goodarzi H, Hosseini SE, Madani H. Adipose-derived mesenchymal stem cells ameliorate lung epithelial injury through mitigating of oxidative stress in mustard lung. Regen Med. 2020 Sep 16. doi: 10.2217/rme-2020-0051. Online ahead of print. PMID 32935623